CLINICAL TRIAL: NCT07011524
Title: A Randomized, Double-blind, Placebo-controlled Phase II Clinical Study Evaluating the Efficacy and Safety of CM512 Injection in Subjects With Moderate-to-severe Asthma.
Brief Title: Study of CM512 Injection in Subjects With Moderate-to-severe Asthma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CM512-103101
Record Dates: First submitted 2025-06-05; First posted 2025-06-08 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental)
  Interventions: Biological: CM512 injection
- Group 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: CM512 injection — subcutaneous injection
  Arms: Group 1
Drug: Placebo — subcutaneous injection
  Arms: Group 2

SUMMARY:
This study is a multicenter, randomized, double-blind, placebo-controlled phase II clinical trial evaluating the efficacy, safety, pharmacokinetics, pharmacodynamics, and immunogenicity of CM512 in subjects with moderate-to-severe asthma.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and comply with procedures of the protocol, and voluntarily sign the Informed Consent Form.
* Age ≥ 18 years old and ≤ 75 years old.
* Body mass index (BMI) ≥ 18.0 kg/(m*m).
* Documented treatment with medium to high dose Inhaled Corticosteroids (ICS) in combination with asthma controller medication for at least 3 months with a stable dose ≥1 month prior to Visit 1.
* Documented history of at least 1 severe asthma exacerbation events within 12 months, and at least one of the exacerbations should occur during the treatment of medium-to-high dose ICS.
* Asthma Control Questionnaire-6 (ACQ-6) score ≥1.5

Exclusion Criteria:

* Women of childbearing potential have a positive pregnancy test result during the screening period; women who are pregnant or lactating.
* With a history of drug abuse within the past 5 years before screening visit.
* Allergic or intolerant to CM512 injection or placebo components, or with a history of severe drug allergies or anaphylactic shock.
* With any medical or non-medical conditions that are not suitable for participation in this study by investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-08-19 (Actual); Primary Completion 2027-07-21 (Estimated); Study Completion 2027-07-21 (Estimated)

PRIMARY OUTCOMES:
Change from the baseline in Forced Expiratory Volume in one second (FEV1) | Up to week 12
  Change from baseline in pre-bronchodilator FEV1 in each dose group at 12 weeks of CM512 treatment compared with placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Ruchong Chen, Principal Investigator — The First Clinical Hospital of Guangzhou Medical University
Locations (1):
- The First Clinical Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China